CLINICAL TRIAL: NCT00253617
Title: Phase III Randomized Study of Double Plastic Endoprosthesis Insertion With Versus Without Adjuvant Photodynamic Therapy Using Porfimer Sodium as Palliative Treatment in Patients With Unresectable Stage III-IV Cholangiocarcinoma
Brief Title: Stent Placement With or Without Photodynamic Therapy Using Porfimer Sodium as Palliative Treatment in Treating Patients With Stage III or Stage IV Cholangiocarcinoma That Cannot Be Removed By Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: AXCAN-PHOCCC04-01; UCLA-0501033-01; CDR0000449701 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2006-12

CONDITIONS: Cholangiocarcinoma of the Extrahepatic Bile Duct; Cholangiocarcinoma of the Gallbladder; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Dihematoporphyrin Ether; Chemotherapy, Adjuvant; Laser Therapy; Photochemotherapy; Phototherapy

INTERVENTIONS:
Drug: porfimer sodium
Procedure: adjuvant therapy
Procedure: laser therapy
Procedure: photodynamic therapy
Procedure: phototherapy

SUMMARY:
RATIONALE: Stent placement may help reduce symptoms caused by the tumor. Photodynamic therapy uses a drug, such as porfimer sodium, that becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed. This may be an effective treatment for cholangiocarcinoma. It is not yet known whether stent placement and photodynamic therapy using porfimer sodium are more effective than stent placement alone in treating cholangiocarcinoma.

PURPOSE: This randomized phase III trial is studying stent placement and photodynamic therapy using porfimer sodium to see how well they work compared to stent placement alone as palliative treatment in treating patients with stage III or stage IV cholangiocarcinoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival time in patients with unresectable Bismuth type III or IV, stage III-IV cholangiocarcinoma treated with double plastic endoprostheses insertion with vs without adjuvant photodynamic therapy using porfimer sodium as palliative treatment.

Secondary

* Compare the effect of these regimens on cholestasis in these patients.
* Compare the 1-year survival rate in patients treated with these regimens.
* Compare health-related quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, controlled, open-label, multicenter study. Patients are stratified according to participating center.

Patients undergo endoscopic or percutaneous drainage followed by insertion of bilateral plastic endoprostheses into the bile ducts. Patients are then randomized to 1 of 2 treatment arms.

* Arm I: Patients receive porfimer sodium IV on day 1. Patients undergo endoscopic laser light therapy to the tumor site on day 3.
* Arm II: Patients receive no further treatment. Quality of life is assessed at baseline and then at weeks 2, 13, 26, 39, 52, and 65.

After completion of study treatment, patients are followed within 30-90 days.

PROJECTED ACCRUAL: A total of 120 patients (60 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed cholangiocarcinoma
* Stage III or IV disease
* Bismuth type III or IV disease
* Tumor mass or stricture on cholangiogram and CT scan
* Unresectable disease

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 30-100%

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 2,000/mm^3
* Platelet count ≥ 50,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Hematocrit ≥ 27%

Hepatic

* PT or INR ≤ 2 times upper limit of normal (correctable with vitamin K)
* No decompensated cirrhosis

Renal

* Not specified

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known porphyria or hypersensitivity to porphyrin
* No clinically significant acute or chronic medial or psychological illness that would preclude study treatment
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or basal cell skin cancer
* No concurrent untreated primary diagnosis of anxiety or depression

PRIOR CONCURRENT THERAPY:

Chemotherapy

* More than 13 weeks since prior and no concurrent chemotherapy

Radiotherapy

* More than 13 weeks since prior and no concurrent brachytherapy or radiotherapy

Surgery

* No prior metal stent insertion
* No prior surgical resection of cholangiocarcinoma

Other

* No prior photodynamic therapy for this disease
* More than 60 days since prior investigational drugs
* No concurrent administration of the following:
* Ursodiol
* Herbal products that may increase bile flow, including any of the following:
* Andrographis paniculata
* Chelidonium majus L
* Curcumin L
* Cynara scolymus L (artichoke)
* Gentiana lutea
* Mentha x piperita (peppermint)
* Peumus boldus Mol
* Taraxacum officinale (dandelion)
* No administration of any of the following within 7 days of porfimer sodium injection:
* Supplements in vitamins C, E, and β-carotene
* Camellia sinensis (green tea)
* Silymarin
* EGb761

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Farrell, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (2):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States
- Axcan Pharma, Incorporated, Mont-Saint-Hilaire, Quebec, Canada